CLINICAL TRIAL: NCT04279418
Title: Effects of Mixed Functional Foods Supplementation on Cognition and Neuroimaging Biomarkers in Adults With Subject Cognitive Decline
Brief Title: Non-pharmacological Intervention for Preclinical Alzheimer's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: XuanwuH 2 (Other)
Responsible Party: Sponsor-Investigator, XuanwuH 2, Professor, Xuanwu Hospital, Beijing
Organization: Xuanwu Hospital, Beijing (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HanYingsc2
Record Dates: First submitted 2020-02-16; First posted 2020-02-21 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Alzheimer Disease; Functional Food; Subjective Cognitive Decline; Intervention; Neuroimaging
Keywords: Subjective cognitive decline; Mixed functional foods; Non-pharmacologic intervention
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mixed functional foods group with SCD (Experimental): Thirty participants in this group will take mixed functional foods for three months.
  Interventions: Dietary Supplement: Mixed functional foods supplementation
- Placebo group with SCD (Placebo Comparator): Thirty participants in this group will take placebo for three months.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Mixed functional foods supplementation — In this project, taking the method of random, double blindness and control, participants in the mixed functional foods group will take functional foods with main compositions of ginsenoside, green tea polyphenols and marine collagen peptide for three months. After that, neuropsychological tests and neuroimaging biomarkers will be compared between functional food group and placebo group.
  Arms: Mixed functional foods group with SCD
Dietary Supplement: Placebo — In this project, taking the method of random, double blindness and control, participants in the placebo group will take placebo for three months. After that, cognitive changes and neuroimaging biomarkers will be compared between functional food group and placebo group.
  Arms: Placebo group with SCD

SUMMARY:
Alzheimer's disease (AD) is the most common form of neurodegenerative disorders leading to dementia. Currently, there has been no effective drugs targeting this disease. Functional food is considered as a potentially non-pharmacologic treatment. In this project, the investigators aim to investigate the effectiveness of a mixed functional food with main compositions of ginsenoside, green tea polyphenols and marine collagen peptide on cognition for individuals with subjective cognitive decline (SCD). Taking the randomized, double-blind, placebo-controlled method, participants in the functional food group will take mixed functional foods for three months and those in the placebo group will take placebo. After that, the investigators will investigate the changes of cognitive function. Furthermore, based on the neuroimaging technique, the regulatory mechanism of functional food in intervening SCD will be revealed from the perspective of altered brain functional activity. In conclusion, these results are beneficial for understanding the therapeutic effect of mixed functional foods as a non-drug treatment for early AD and further elucidating the potential brain mechanism, which are of great values in solving scientific and clinical practice issues.

DETAILED DESCRIPTION:
Currently, there has been no effective therapy for Alzheimer's disease (AD). Functional food is now considered as a potentially non-pharmacologic intervention and supplementation of functional food may positively affect cognitive function for patients with AD. However, there are few existing studies involving the role of mixed functional foods with multiple compositions on cognition and neuroimaging biomarkers for subjective cognitive decline (SCD).

Sixty participants with SCD will be recruited in this three-month, randomized, double-blind, placebo-controlled trial. Each group had thirty participants. Participants in the functional food group will take mixed functional foods for three months and those in the placebo group will take placebo. After that, the investigators will investigate the changes of memory measures, which is the primary outcome. Furthermore, based on the neuroimaging technique of functional near-infrared spectroscopy (fNIRS), the regulatory mechanism of mixed functional foods in intervening SCD will be revealed from the perspective of altered brain functional activity.

In conclusion, these results are beneficial for understanding the therapeutic effect of mixed functional foods as a non-drug therapy for preclinical AD and further elucidating the potential brain mechanism, which are of great values in solving scientific and clinical practice issues.

ELIGIBILITY:
Inclusion Criteria:

* 50-79 years old, right-handed and Mandarin-speaking subjects;
* self-experienced persistent decline in cognitive capacity in comparison with a previously normal status and unrelated to an acute event;
* normal age-adjusted, gender-adjusted and education-adjusted performance on standardised cognitive tests;
* concerns (worries) associated with memory complaint;
* failure to meet the criteria for MCI or dementia

Exclusion Criteria:

* a history of stroke;
* major depression (Hamilton Depression Rating Scale score > 24 points);
* other central nervous system diseases that may cause cognitive impairment, such as Parkinson's disease, tumors, encephalitis and epilepsy;
* cognitive impairment caused by traumatic brain injury;
* systemic diseases, such as thyroid dysfunction, syphilis and HIV;
* a history of psychosis or congenital mental growth retardation.

Ages: 50 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Changes of Auditory Verbal Learning Test (AVLT) score | Three months
  After intervention for three months, the investigators will compare memory changes based on Auditory Verbal Learning Test (AVLT) scale in two groups, in order to investigate the therapeutic effectiveness of mixed functional foods supplementation. The scale of AVLT focuses on the memory domain, especially AVLT-long delayed memory, with cut-off points as 5 (50-59 years old), 4 (60-69 years old), 3 (70-79 years old) and AVLT-recognition, with cut-off points as 20 (50-59 years old), 19 (60-69 years old), 18 (70-79 years old). Higher scores mean a better outcome.

SECONDARY OUTCOMES:
FNIRS-based brain functional activity changes | Three months
  At baseline and post-intervention visits, the brain functional activity data will be collected using functional near-infrared spectroscopy (fNIRS) technique. The investigators will compare the changes of brain functional activity based on the measure of oxyhemoglobin concentration signal with relatively high signal to noise ratio (SNR) in two groups, in order to reveal the regulatory mechanism of mixed functional foods in intervening SCD persons.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Han, PhD, Principal Investigator — Xuanwu Hospital of Capital Medical University
Locations (1):
- Department of Neurolgy, Xuanwu Hospital of Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The information of neuropsychological tests, neuroimaging data are to be shared with other researchers.
Supporting Information: Study Protocol
Time Frame: When summary data are published or starting 6 months after publication.
Access Criteria: The information of neuropsychological tests, neuroimaging data will be shared.